CLINICAL TRIAL: NCT00766636
Title: A Randomized Phase II Study of Preoperative Chemotherapy (Gemcitabine and Erlotinib) With or Without Radiation Therapy for Patients With Resectable Adenocarcinoma of the Pancreas
Brief Title: Preoperative Chemotherapy (Gemcitabine and Erlotinib) With or Without Radiation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0459
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-08

CONDITIONS: Pancreatic Cancer
Keywords: Adenocarcinoma of the pancreatic head; Pancreaticoduodenectomy; Preoperative chemotherapy; Chemoradiation; Resectable pancreatic cancer; Surgical removal of the pancreas and duodenum; External-beam radiation therapy; EBRT; Gemcitabine; Erlotinib
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiotherapy; Erlotinib Hydrochloride; Surgical Procedures, Operative; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine + Erlotinib Without Radiation (Experimental): Gemcitabine + Erlotinib without radiation - Arm A: Gemcitabine 1000 mg/M^2 given intravenously over 100 min. every week for 6 doses beginning day 1 (days 1, 8, 15, 22, 29, 36) +/- 1 day. Erlotinib 100 mg daily by mouth on days 1-42.
  Surgical removal of the pancreas and duodenum.
  Interventions: Drug: Gemcitabine; Drug: Erlotinib; Procedure: Surgery
- Gemcitabine + Erlotinib With Radiation (Experimental): Gemcitabine + Erlotinib with radiation - Arm B: Gemcitabine 400 mg/M^2 given intravenously over 40 min. every week for 6 doses beginning day 1 (days 1, 8, 15, 22, 29, 36) +/- 1 day. Erlotinib 100 mg daily by mouth on days 1-42. Radiation therapy 1 time each day for 5 days in a row for 5 1/2 weeks starting on Day 1 for a total of 50.4 Gy. Surgical removal of the pancreas and duodenum.
  Interventions: Drug: Gemcitabine; Radiation: Radiation Therapy; Drug: Erlotinib; Procedure: Surgery

INTERVENTIONS:
Drug: Gemcitabine — Arm A:
  1000 mg/M^2 given intravenously over 100 min. every week for 6 doses beginning day 1 (days 1, 8, 15, 22, 29, 36) +/- 1 day.
  Arm B:
  400 mg/M^2 given intravenously over 40 min. every week for 6 doses beginning day 1 (days 1, 8, 15, 22, 29, 36) +/- 1 day.
  Other Names: Gemzar
Radiation: Radiation Therapy — 1 time each day for 5 days in a row for 5 1/2 weeks starting on Day 1 for a total of 50.4 Gy.
  Other Names: RT; Radiotherapy; External Beam Radiation Therapy; EBRT
  Arms: Gemcitabine + Erlotinib With Radiation
Drug: Erlotinib — 100 mg daily by mouth on days 1-42.
  Other Names: Erlotinib Hydrochloride; OSI-774; Tarceva
Procedure: Surgery — Surgical removal of the pancreas and duodenum
  Other Names: pancreaticoduodenectomy; resection

SUMMARY:
Primary Objective:

To assess margin positive resection rate (R1 resection rate; defined as "tumor within 2 mm of surgical margin on final pathology report") in patients treated with preoperative chemotherapy (gemcitabine and erlotinib) with or without external-beam radiation therapy followed by pancreaticoduodenectomy for adenocarcinoma of the pancreatic head.

Secondary Objectives:

* To assess disease free survival
* To assess overall survival
* To assess patterns of local and distant failure

DETAILED DESCRIPTION:
The Study Drugs:

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die.

Erlotinib is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Screening Tests:

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* You will have a complete physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests. This routine blood draw will include a pregnancy test for women who are able to have children. To take part in this study, the pregnancy test must be negative.
* You will be asked about any side effects you may have experienced.
* Urine will be collected for routine tests.
* You will have chest x-rays and computed tomography (CT) scans of the abdomen to check the status of the disease.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to receive either chemotherapy without radiation (Group A) or chemotherapy with radiation (Group B). You will have an equal chance of being in either group.

Pre-Surgery Study Drug Administration:

* If you are in Group A, you will receive gemcitabine over about 90 minutes 1 time each week (Days 1, 8, 15, 22, 29, 36 [+/- 2 Days]. You will take erlotinib by mouth, with water, 1 hour before eating or 2 hours after eating 1 time daily on Days 1-42.
* If you are in Group B, you will receive gemcitabine over about 40 minutes 1 time each week (Days 1, 8, 15, 22, 29, 36, [+/- 2 Days]). You will take erlotinib by mouth, with water, 1 hour before eating or 2 hours after eating 1 time daily on Days 1-42. You will also receive radiation therapy 1 time each day for 5 days in a row (Monday through Friday) for 5 1/2 weeks starting on Day 1. You will sign a separate consent form for the radiation therapy. If any days of radiation therapy are missed, you will make up the missed day(s) at the end of therapy so you receive the full amount of radiation therapy.

Post-Surgery Study Drug Administration:

For all participants, starting within 12 weeks after the surgery, you will receive gemcitabine over 100 minutes on Days 1, 8, and 15 [+/- 2 Days]) of each 4 weeks cycle. You will also take erlotinib by mouth with water 1 hour before eating or 2 hours after eating 1 time daily for 4 weeks.

You may be able to receive your postoperative therapy closer to home by an outside cancer doctor. This will be up to the treating cancer doctor at M. D. Anderson. A research nurse will contact you at least every other week by telephone. Participants who need radiation treatment will only be allowed to receive radiation treatment at M. D. Anderson Cancer Center.

Surgery:

All participants will have chest x-rays and CT scans performed approximately 4 weeks after the last dose of the study drug combination to check the status of the disease. If the disease has not gotten worse, and the study doctor thinks it is in your best interest, you will be scheduled to have surgery to remove the pancreas and duodenum. You will sign a separate consent form for the surgery.

If you are not found to be eligible for surgery, your participation on this study end at this time.

Length of Study:

You will be taken off study early if the disease gets worse, you experience intolerable side effects, or the study doctor thinks it is no longer in your best interest to continue to receive the study drug. You will remain on the study for approximately 10 months.

Follow-Up Visit:

After your participation on this study is complete, you will have a chest x-ray and a CT scan every 4 months for 2 years.

This is an investigational study. Gemcitabine and Erlotinib are both FDA and commercially available, but their use together with radiation therapy is investigational.

Up to 190 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic proof of adenocarcinoma of the pancreatic head or uncinate process is required prior to treatment. Islet cell tumors are not eligible.
2. Patients must be staged with a physical exam, CXR, and contrast-enhanced CT. Only potentially resectable patients are eligible. Potentially resectable defined as: a) no extra pancreatic disease, b) no evidence (on CT) of tumor extension to the celiac axis or SMA, and c) no evidence (CT or angiogram) of occlusion of the SMV or SMPV confluence. Visceral angiography is optional. Laparoscopic staging is not part of the pretreatment evaluation for this study. Laparoscopy may be performed prior to planned laparotomy at surgeon's discretion. Staging needs to be done within 28 days of enrollment.
3. Patients cannot have known hepatic or peritoneal metastases detected by ultrasound (US), CT scan, or laparotomy prior to treatment
4. There will be no upper age restriction; patients with Karnofsky performance status greater than 70 are eligible.
5. Adequate renal, and bone marrow function: • Leukocytes >= 3,000/uL • Absolute neutrophil count >= 1,500/uL • Platelets >= 100,000/Ul • Serum creatinine <= 2.0 mg/dL
6. Hepatic function (endoscopic or percutaneous drainage as needed) • Total bilirubin < = 2 X institutional upper limits of normal (ULN) • AST (SGOT)/ALT (SGPT) <= 5 X institutional ULN
7. Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude protocol therapy.
8. Pregnant women with a positive (blood B-HCG) pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to practice adequate contraception and to refrain from breast feeding, as specified in the informed consent.
9. Patients must sign a study-specific consent form, which is attached to this protocol.

Exclusion Criteria:

1. Tumors in the body or tail of the pancreas (to the left of the portal -SMV confluence) are not eligible.
2. Unstable angina or New York Heart Association (NYHA) Grade II or greater congestive heart failure
3. Known presence of central nervous system or brain metastases
4. Inability to comply with study and/or follow-up procedures
5. Patients < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-09; Primary Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason B. Fleming, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 4, 2008 to December 7, 2009. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 5 participants enrolled, one withdrew consent and the others did not complete treatment.
Period: Overall Study
Arm/Group | Gemcitabine + Erlotinib Without Radiation | Gemcitabine + Erlotinib With Radiation
Started | 3 | 2
Completed | 0 (Number that completed pre- and post-operative therapy as well as surgery.) | 0
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Incomplete Treatment | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant in Gemcitabine + Erlotinib with Radiation did not receive any treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine + Erlotinib Without Radiation | Gemcitabine + Erlotinib With Radiation | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 61 [44 to 63] | 67.5 [64 to 71] | 63 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Difference in Positive Margin Resection (R1) Rate in Patients Undergo Surgery Between the Two Treatment Groups.
Description: Difference in positive margin resection (R1) rate in patients who undergo surgery between the two treatment groups. Margin resection rate is defined as number of patients with R1 margin divided by the total number of patients who received surgery in that arm. Eligible patients will be equally (1:1 ratio) randomized to one of the two arms to receive either Gemcitabine and Erlotinib or Gemcitabine and Erlotinib and radiation as preoperative therapy. Surgery to be performed approximately 4 weeks after preoperative therapy. R1 resection defined as as tumor within 2mm of the surgical margin on the final pathology report
Time Frame: Following resection performed at time of surgery, day 36 of treatment +/- 5 days
Population: The study was terminated early without enough patients to perform any analysis between the groups. Of the five registered, one withdrew prior to any treatment and the others either had disease progression or left prior to surgery with incomplete preoperative regimen.
Arm/Group | Gemcitabine + Erlotinib Without Radiation | Gemcitabine + Erlotinib With Radiation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed from the time of consent until two years following surgery. Collection Period: September 2008 to April 2011.
Arm/Group | Gemcitabine + Erlotinib Without Radiation | Gemcitabine + Erlotinib With Radiation
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Erlotinib Without Radiation (N=3) | Gemcitabine + Erlotinib With Radiation (N=2)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes